CLINICAL TRIAL: NCT00184743
Title: Investigation of the Efficacy and Safety of NN-220 for 48 Weeks in Adults With Growth Hormone Deficiency
Brief Title: Long-term Trial on Growth Hormone Deficiency in Adults (GHDA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHLIQUID-1519; JapicCTI-050133 (Registry Identifier: japic)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Japan. To investigate the long-term efficacy as assessed by change in fat mass and safety after 48 weeks of treatment of Growth Hormone in adults with Growth Hormone Deficiency, comparing two different treatment regiments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed GHLiquid-1518.
* If the subject has a history of treatment for a tumor of pituitary or peripheral site, two years or more have to be passed since completion of surgery, radiotherapy or other treatment, and recurrence of the underlying disease to be excluded.
* Appropriate replacement therapy has been administered for more than 24 weeks for the treatment of other pituitary hormone deficiencies.

Exclusion Criteria:

* Subject with a history of acromegaly.
* Subject with diabetes mellitus.
* Subject suffering from malignancy.
* Several medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2003-12-06 (Actual); Primary Completion 2005-12-28 (Actual); Study Completion 2005-12-28 (Actual)

PRIMARY OUTCOMES:
Percent change in truncal fat (kg) | from the baseline to the end of treatment

SECONDARY OUTCOMES:
Adverse events
Change in Total body fat, Total LBM, etc. from the baseline to the end of treatment
Lipid-related laboratory tests (total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglyceride)
FPG, insulin, and HbA1C
IGF-I SDS, IGFBP-3 SDS, and IGF-I/IGFBP-3 molar ratio
Clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Derived] Chihara K, Kato Y, Shimatsu A, Tanaka T, Kohno H. Efficacy and safety of individualized growth hormone treatment in adult Japanese patients with growth hormone deficiency. Growth Horm IGF Res. 2008 Oct;18(5):394-403. doi: 10.1016/j.ghir.2008.02.002. Epub 2008 Apr 18. PMID 18395480
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com